CLINICAL TRIAL: NCT01811732
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active-controlled Study to Evaluate the Efficacy and Safety of Delafloxacin Compared With Vancomycin + Aztreonam in Patients With Acute Bacterial Skin and Skin Structure Infections
Brief Title: Delafloxacin Versus Vancomycin and Aztreonam for the Treatment of Acute Bacterial Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RX-3341-302; 2012-001767-71 (EudraCT Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-15 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections
Keywords: Bacterial skin infection; skin infection; infection; skin; delafloxacin; vancomycin; aztreonam; MRSA bacteria; bacterial infection; Anti-Infective Agents; Anti-Bacterial Agents
MeSH Terms: conditions — Skin Diseases, Bacterial; Cellulitis; Infections; Bacterial Infections | interventions — delafloxacin; Vancomycin; Aztreonam; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delafloxacin plus placebo (Experimental): Delafloxacin 300 mg IV every 12 hours for a minimum of 10 and up to a maximum of 28 doses
  Interventions: Drug: Delafloxacin; Drug: Placebo
- Vancomycin plus Aztreonam + placebo (Active Comparator): Vancomycin 15 mg/kg IV plus two grams Aztreonam every 12 hours for a minimum of 10 and up to a maximum of 28 doses (Aztreonam was discontinued as soon as possible if a gram-negative organism was not identified in baseline cultures)
  Interventions: Drug: Vancomycin; Drug: Aztreonam; Drug: Placebo

INTERVENTIONS:
Drug: Delafloxacin — Delafloxacin
  Other Names: RX-3341
  Arms: Delafloxacin plus placebo
Drug: Vancomycin — Vancomycin
  Arms: Vancomycin plus Aztreonam + placebo
Drug: Aztreonam — Aztreonam
  Arms: Vancomycin plus Aztreonam + placebo
Drug: Placebo — Placebo
  Other Names: 5% Dextrose; D5W

SUMMARY:
This study was designed to evaluate the efficacy of delafloxacin patients with acute bacterial skin and soft tissue infections (ABSSSI).

DETAILED DESCRIPTION:
The efficacy and safety of delafloxacin, compared to that of vancomycin plus aztreonam, will be evaluated in a population of patients with acute bacterial skin and soft tissue infections (ABSSSI), including major cutaneous abscesses, wound infections, cellulitis/erysipelas, and burn-related infections.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) men or women with a diagnosis of Acute Bacterial Skin and Skin Structure Infections (ABSSSI) (cellulitis/erysipelas, wound infection, major cutaneous abscess, or burn infection) with surrounding redness of a minimum surface area of 75 cm^2 and at least two signs of systemic infection
* In the opinion of the investigator, the subject must require and be a suitable candidate for IV antibiotic therapy, and the subject must be able and willing to comply with protocol requirements

Exclusion Criteria:

* A medical history of significant hypersensitivity or allergic reaction to quinolones, beta-lactams, vancomycin, or vancomycin derivatives according to the judgment of the investigator
* Women who are pregnant or lactating
* Any chronic or underlying skin condition at the site of infection that may complicate the assessment of response, including infection involving a prosthetic joint, human or animal bite, osteomyelitis, decubitus ulcer, diabetic foot ulcer, septic arthritis, mediastinitis, necrotizing fasciitis, anaerobic cellulitis, or synergistic necrotizing cellulitis, myositis, tendinitis, endocarditis, sustained shock, gangrene or gas gangrene; burns covering ≥10% of body surface area; severely impaired arterial blood supply to an extremity with an ABSSSI, deep vein thrombosis or superficial thrombophlebitis, and requiring either an amputation or multiple debridement procedures
* Receipt of systemic antibiotic therapy in the 14 days before enrollment unless 1 of the following was documented:

  1. Received ≥ 48 hours of antibiotic therapy for ABSSSI AND clinical progression is documented (i.e., not by patient history alone).
  2. Recently (within 14 days) completed a treatment course with an antibacterial drug for an infection other than ABSSSI and the drug does not have activity against bacterial pathogens that cause ABSSSI.
  3. Received only 1 dose of either a single, potentially effective, short-acting antimicrobial drug or drug regimen for ABSSSI.
* Any underlying disease that, in the opinion of the investigator, could interfere with the subject's ability to participate in the study including severe cardiac disease, known history of liver disease, end-stage renal disease, malignancy, psychiatric disorder, ongoing treatment for seizures or untreated history of seizures, or life expectancy of <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue K. Cammarata, MD, Study Director — Melinta Therapeutics, Inc.
Locations (44):
- United States (17):
  - Melinta Investigational Site, Montgomery, Alabama
  - Melinta Investigational Site, Anaheim, California
  - Melinta Investigational Site, Chula Vista, California
  - Melinta Investigational Site, La Mesa, California
  - Melinta Investigational Site, Long Beach, California
  - Melinta Investigational Site, Los Angeles, California
  - Melinta Investigational Site, Modesto, California
  - Melinta Investigational Site, Oceanside, California
  - Melinta Investigational Site, Pasadena, California
  - Melinta Investigational Site, Stockton, California
  - Melinta Investigational Site, Miramar, Florida
  - Melinta Investigational Site, Minneapolis, Minnesota
  - Melinta Investigational Site, Butte, Montana
  - Melinta Investigational Site, Las Vegas, Nevada
  - Melinta Investigational Site, Somers Point, New Jersey
  - Melinta Investigational Site, Smyrna, Tennessee
  - Melinta Investigational Site, Richmond, Texas
- Croatia (2):
  - Melinta Investigational Site, Slavonski Brod
  - Melinta Investigational Site, Zagreb
- Israel (5):
  - Melinta Investigational Site, Haifa
  - Melinta Investigational Site, Kfar Saba
  - Melinta Investigational Site, Nazareth
  - Melinta Investigational Site, Safed
  - Melinta Investigational Site, Tel Aviv
- Latvia (4):
  - Melinta Investigational Site, Daugavpils
  - Melinta Investigational Site, Liepāja
  - Melinta Investigational Site, Riga
  - Melinta Investigational Site, Valmiera
- Russia (4):
  - Melinta Investigational Site, Moscow
  - Melinta Investigational Site, Perm
  - Melinta Investigational Site, Saint Petersberg
  - Melinta Investigational Site, Vsevolozhsk
- Spain (4):
  - Melinta Investigational Site, Barcelona
  - Melinta Investigational Site, Granada
  - Melinta Investigational Site, Málaga
  - Melinta Investigational Site, Valencia
- Ukraine (8):
  - Melinta Investigational Site, Chemivtsi
  - Melinta Investigational Site, Cherkasy
  - Melinta Investigational Site, Dnipropetrovsk
  - Melinta Investigational Site, Ivano-Frankivsk
  - Melinta Investigational Site, Klarkiv
  - Melinta Investigational Site, Lviv
  - Melinta Investigational Site, Odesa
  - Melinta Investigational Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lodise T, Corey R, Hooper D, Cammarata S. Safety of Delafloxacin: Focus on Adverse Events of Special Interest. Open Forum Infect Dis. 2018 Sep 10;5(10):ofy220. doi: 10.1093/ofid/ofy220. eCollection 2018 Oct. PMID 30349845
- [Derived] Pullman J, Gardovskis J, Farley B, Sun E, Quintas M, Lawrence L, Ling R, Cammarata S; PROCEED Study Group. Efficacy and safety of delafloxacin compared with vancomycin plus aztreonam for acute bacterial skin and skin structure infections: a Phase 3, double-blind, randomized study. J Antimicrob Chemother. 2017 Dec 1;72(12):3471-3480. doi: 10.1093/jac/dkx329. PMID 29029278
- [Derived] McCurdy S, Lawrence L, Quintas M, Woosley L, Flamm R, Tseng C, Cammarata S. In Vitro Activity of Delafloxacin and Microbiological Response against Fluoroquinolone-Susceptible and Nonsusceptible Staphylococcus aureus Isolates from Two Phase 3 Studies of Acute Bacterial Skin and Skin Structure Infections. Antimicrob Agents Chemother. 2017 Aug 24;61(9):e00772-17. doi: 10.1128/AAC.00772-17. Print 2017 Sep. PMID 28630189

RESULTS

PARTICIPANT FLOW:
Groups:
- Delafloxacin Plus Placebo: 300 mg IV every 12 hours, for a minimum of 10 and up to a maximum of 28 doses
  Delafloxacin: Delafloxacin
  Placebo: Placebo
- Vancomycin Plus Aztreonam + Placebo: Vancomycin 15 mg/kg IV plus two grams Aztreonam every 12 hours for a minimum of 10 and up to a maximum of 28 doses
  Vancomycin: Vancomycin
  Aztreonam: Aztreonam
  Placebo: Placebo
Period: Overall Study
Arm/Group | Delafloxacin Plus Placebo | Vancomycin Plus Aztreonam + Placebo
Started | 331 | 329
Completed (Completed the Late Follow-Up (LFU) Visit) | 276 | 271
Not Completed | 55 | 58
Not completed — Lost to Follow-up | 24 | 30
Not completed — Withdrawal by Subject | 16 | 10
Not completed — Adverse Event | 3 | 9
Not completed — Lack of Efficacy | 3 | 1
Not completed — Non-compliance with study drug/procedure | 3 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Death | 1 | 1
Not completed — Insufficient venous access | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Subject incarcerated | 1 | 2
Not completed — Admitted to another facility | 1 | 0
Not completed — Correct study drug not available on site | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all patients who were randomly assigned to treatment.
Groups:
- Delafloxacin + Placebo: 300mg iv every 12 hours for a minimum of 10 and up to a maximum of 28 doses
  Delafloxacin: Delafloxacin
  Placebo: Placebo
- Vancomycin Plus Aztreonam + Placebo: Vancomycin 15mg/kg iv plus two grams Aztreonam every 12 hours for a minimum of 10 and up to a maximum of 28 doses
  Vancomycin: Vancomycin
  Aztreonam: Aztreonam
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Delafloxacin + Placebo | Vancomycin Plus Aztreonam + Placebo | Total
Number analyzed (Participants) | 331 | 329 | 660
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.91) | 45.3 (14.44) | 45.8 (14.18)
Age, Customized [Count of Participants; unit: Participants]
  <= 65 years | 309 | 309 | 618
  > 65 years | 22 | 20 | 42
  > 75 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 120 | 245
  Male | 206 | 209 | 415
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 103 | 204
  Not Hispanic or Latino | 230 | 226 | 456
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 27 | 19 | 46
  White | 297 | 304 | 601
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 268 | 274 | 542
  Europe | 63 | 55 | 118
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m2] | 28.36 (6.423) | 27.86 (6.363) | 28.11 (6.393)
BMI ranges [Count of Participants; unit: Participants]
  < 25 | 113 | 125 | 238
  >= 25 | 218 | 204 | 422
  >= 30 | 120 | 94 | 214
  >= 35 | 53 | 42 | 95
Presence of Diabetes [Count of Participants; unit: Participants] | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Objective Response at 48 to 72 Hours (FDA Primary Endpoint)
Description: A patient was considered a responder if s/he had a ≥20% reduction in size of the area of erythema associated with the baseline ABSSSI, as determined by digital planimetry of the leading edge and had none of the reasons for clinical failure; a patient was considered a non-responder (failure) if s/he had <20% reduction in size of the area of erythema associated with the baseline ABSSSI as determined by digital planimetry of the leading edge, or had major intervention such as another antibiotic or surgical intervention or died within 74 hours after initiation of study drug.
Time Frame: 48 to 72 hours after starting treatment
Population: ITT Population
Measure: Count of Participants; unit: Participants
Groups:
- Delafloxacin Plus Placebo: 300mg iv every 12 hours for a minimum of 10 and up to a maximum of 28 doses
  Delafloxacin: Delafloxacin
  Placebo: Placebo
Arm/Group | Delafloxacin Plus Placebo | Vancomycin Plus Aztreonam + Placebo
Number analyzed (Participants) | 331 | 329
Participants
  Responder | 259 | 266
  Non-Responder | 72 | 63
Statistical Analysis 1: Comparison: Delafloxacin Plus Placebo vs Vancomycin Plus Aztreonam + Placebo; Test type: Non-Inferiority — A 2-sided 95% confidence interval (CI) for noninferiority testing was computed based on the difference in sample rates for vancomycin + aztreonam and delafloxacin at the primary endpoint. If the upper limit (UL) of the CI was less than 0.10, delafloxacin would be considered noninferior to vancomycin + aztreonam; Difference in Responder Rates = -2.6, 95% CI 2-sided [-8.8 to 3.6]

2. Secondary Outcome: Investigator Assessment at the Follow-up Visit (EMA Primary Endpoint)
Description: A patient was considered a Cure if all baseline signs and symptoms of ABSSSI had resolved; if some symptoms remained, but the patient was improved to the extent that no additional antibiotic treatment was necessary, the response was Improved. A patient was considered a Failure for any of the following reasons: nonstudy antibacterial drug therapy was required because of lack of efficacy after at least 4 doses of study drug or for a treatment-related AE; study antibacterial drug therapy was required for longer than 28 doses; and/or unplanned surgical intervention was needed after study entry except for limited bedside debridement and standard wound care. Improved and Indeterminate responses were considered failures in the primary analysis.
  A sensitivity analysis was also performed, in which the assigned responses were Success (Cure + Improved) or Failure (Failure + Indeterminate/Missing).
Time Frame: Study Day 14 +/- 1 day
Population: ITT Population
Measure: Count of Participants; unit: Participants
Groups:
- Delafloxacin Plus Placebo: 300mg iv every 12 hours, for a minimum of 10 and up to a maximum of 28 doses
  Delafloxacin: Delafloxacin
  Placebo: Placebo
Arm/Group | Delafloxacin Plus Placebo | Vancomycin Plus Aztreonam + Placebo
Number analyzed (Participants) | 331 | 329
Participants
  Cure | 172 | 166
  Improved | 98 | 108
  Failure | 9 | 7
  Indeterminate | 52 | 48

3. Secondary Outcome: Investigator Assessment at the Late Follow-up Visit
Description: as for outcome 2
Time Frame: Study Day 21 to 28
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin Plus Placebo | Vancomycin Plus Aztreonam + Placebo
Number analyzed (Participants) | 331 | 329
Participants
  Cure | 233 | 219
  Improved | 32 | 48
  Failure | 9 | 6
  Indeterminate/Missing | 57 | 56

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the patient signed the ICF through the follow-up telephone contact 30 days after the last dose of study drug (up to 45 days).
Description: AE data are only included for the safety population which included all patients in the ITT population who received at least 1 dose of study drug.
Arm/Group | Delafloxacin Plus Placebo | Vancomycin Plus Aztreonam + Placebo
All-Cause Mortality (participants affected / at risk) | 1/324 | 1/326
Serious Adverse Events (participants affected / at risk) | 12/324 | 12/326
Other Adverse Events (participants affected / at risk) | 91/324 | 111/326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delafloxacin Plus Placebo (N=324) | Vancomycin Plus Aztreonam + Placebo (N=326)
Cellulitis (Infections and infestations) | 2 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Peritonitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Polysubstance dependence (Psychiatric disorders) | 1 | 0
Substance-induced mood disorder (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Peripheral ischemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delafloxacin Plus Placebo (N=324) | Vancomycin Plus Aztreonam + Placebo (N=326)
Infection (Infections and infestations) | 28 | 25
Infusion site extravasation (General disorders) | 28 | 44
Diarrhea (Gastrointestinal disorders) | 27 | 10
Nausea (Gastrointestinal disorders) | 24 | 28
Headache (Nervous system disorders) | 10 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Melinta has the right to first publication of results, which would be made in conjunction with the PIs from all appropriate sites. Thereafter, PIs may publish results provided the PI submits the proposed publication to Melinta for review at least 60 days prior to the date of the proposed publication. Melinta may remove any information that is considered confidential and/or proprietary. If a publication is not submitted within 12 months of study conclusion, the PI may publish results.